CLINICAL TRIAL: NCT02820935
Title: A Phase 1, Open-label, Single-center Study to Evaluate the Effect of Cytochrome P450 (CYP) 3A Inhibition and Induction on the Pharmacokinetics of CC-220 in Healthy Subjects
Brief Title: Study to Evaluate the Effect of Cytochrome P450 (CYP) 3A Inhibition and Induction on the Pharmacokinetics of CC-220 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CC-220-CP-003
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Pharmacokinetics
Keywords: Cytochrome P450; Pharmacokinetics; CC-220; Healthy Subjects
MeSH Terms: interventions — iberdomide; Rifampin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1, Period 1: CC-220 (Experimental): Single dose of 0.6mg CC-220
  Interventions: Drug: CC-220
- Part 1, Period 2: itraconazole with CC-220 (Experimental): Multiple does of 200 mg itraconazole alone, with a single dose of 0.6 mg CC-220 plus itraconazole
  Interventions: Drug: CC-220; Drug: Itraconazole
- Part 2, Period 1: CC-220 (Experimental): Single dose of 0.6mg CC-220
  Interventions: Drug: CC-220
- Part 2, Period 2: rifampin with CC-220 (Experimental): Multiple doses of 600 mg rifampin alone, with a single dose of 0.6 mg CC-220 plus rifampin
  Interventions: Drug: CC-220; Drug: Rifampin

INTERVENTIONS:
Drug: CC-220
Drug: Rifampin
  Arms: Part 2, Period 2: rifampin with CC-220
Drug: Itraconazole
  Arms: Part 1, Period 2: itraconazole with CC-220

SUMMARY:
This is a two-part study to be conducted at a single study site in the US. Both parts of the study may be conducted in parallel.

A total of approximately 38 subjects will participate in this study, with approximately 19 subjects in Part 1 and approximately 19 subjects in Part 2. Each subject may only participate in one of the parts.

DETAILED DESCRIPTION:
This is a two part study to be conducted at a single study site. Both parts of the study may be conducted in parallel.

A total of approximately 38 subjects will participate in this study, with approximately 19 subjects in Part 1 and approximately 19 subjects in Part 2. Each subject may only participate in one of the parts.

Each Part will consist of 2 study periods. Part 1 and Part 2, each subject will participate in a Screening phase, one baseline visit per period, one dosing phase per period, and follow-up telephone call.

In Part 1, subjects will receive a single dose of CC-220 in Period 1 and, following an appropriate washout, multiple doses of itraconazole plus one dose of itraconazole with CC-220 in Period 2. In Part 2, subjects will receive CC-220 in Period 1 and, following an appropriate washout, multiple doses of rifampin plus one dose of rifampin with CC-220 in Period 2.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 and ≤ 65 years of age at the time of signing the informed consent form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject is in good health as determined by a Physical examination (PE) at screening.
5. Subject agrees to abide by the requirements and restrictions outlined in the CC-220 Pregnancy Prevention Plan for Subjects in Clinical Trials.
6. Female subjects not of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a follicle-stimulating hormone [FSH] level of > 40 IU/L at screening).
7. Male subjects must:

   a. Practice true abstinence1 (which must be reviewed on a monthly basis and source documented) or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or female of childbearing potential (FCBP)2 while participating in the study, during dose interruptions, and for at least 28 days after the last dose of investigational Product (IP), even if he has undergone a successful vasectomy.
8. Subject has body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.

1 True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception). 2 A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point; 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).

9. Subject has clinical laboratory safety test results that are within normal limits or acceptable to the Investigator. Platelet count, absolute neutrophil count, and absolute lymphocyte count must be above the lower limit of normal at screening.

10. Subject is afebrile, with supine systolic blood pressure (BP) ≥ 90 and ≤ 140 mmHg, supine diastolic BP ≥ 50 and ≤ 90 mmHg, and pulse rate ≥ 40 and ≤ 110 bpm at screening.

11. Subject has a normal or clinically acceptable 12-lead ECG (Electrocardiogram) at screening. In addition:

1. If male, subject has a corrected QT value (based on Fridericia's formula) ≤ 430 msec at screening.
2. If female, subject has a corrected QT value (based on Fridericia's formula) ≤ 450 msec at screening.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant and relevant medical condition (including but not limited to neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders), laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject is a female of childbearing potential, pregnant, or breastfeeding.
5. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or five half-lives of that investigational drug, if known (whichever is longer).
6. Subject has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days prior to the first dose administration.
7. Subject has used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days prior to the first dose administration.
8. Subject has used CYP3A inducers and/or inhibitors (including St. John's wort) within 30 days prior to the first dose administration. The Indiana University "Cytochrome P450 Drug Interaction Table" should be utilized to determine inhibitors and/or inducers of CYP3A.
9. Subject has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion, eg, bariatric procedure. Appendectomy and cholecystectomy are acceptable.
10. Subject donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
11. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before the first dose administration, or positive drug screening test reflecting consumption of illicit drugs.
12. Subject has a history of alcohol abuse (as defined by the current version of the Diagnostic and Statistical Manual (DSM)) within 2 years before the first dose administration, or positive alcohol screen.
13. Subject is known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.
14. Subject smokes > 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
15. Subject is part of the clinical staff personnel or a family member of the clinical site staff.
16. Subject has received immunization with a live or live attenuated vaccine within 2 months prior to administration of the first dose of IP or is planning to receive immunization with a live or live attenuated vaccine for 2 months after administration of the last dose of Investigational Product (IP).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics- Cmax | Up to 96 hours
  Maximum plasma concentration
Pharmacokinetics- AUC∞ | Up to 96 hours
  Area under the plasma concentration from time zero extrapolated to infinity

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 2 month
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Maria Palmisano, MD, Study Director — Celgene Corporation
Locations (1):
- PPD Development, LP, Austin, Texas, United States

REFERENCES:
- [Derived] Gaudy A, Atsriku C, Ye Y, MacGorman K, Liu L, Xue Y, Surapaneni S, Palmisano M. Evaluation of iberdomide and cytochrome p450 drug-drug interaction potential in vitro and in a phase 1 study in healthy subjects. Eur J Clin Pharmacol. 2021 Feb;77(2):223-231. doi: 10.1007/s00228-020-03004-w. Epub 2020 Sep 23. PMID 32965548